CLINICAL TRIAL: NCT00420069
Title: Biphasic Extrathoracic Cuirass Ventilation During Dental Treatment Under Deep Sedation
Brief Title: Biphasic Extrathoracic Cuirass Ventilation During Dental Treatment
Status: Withdrawn | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: di123HMO-CTIL
Record Dates: First submitted 2007-01-07; First posted 2007-01-09 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2007-01

CONDITIONS: Blood Gas Monitoring, Transcutaneous

INTERVENTIONS:
Device: MRTX device — device for ventilation

SUMMARY:
The MRTX portable lightweight respirator (MRTX) provides noninvasive respiratory support using biphasic extrathoracic ventilation via a cuirass fitted around the patient's chest.The aim of the study is to evaluate the efficacy of the MRTX during dental treatment under deep sedation in comparison with the conventional treatment where children are only under monitor and only intervention is done when required.Twenty healthy children (ASA1) will wear the cuirass. PO2 saturation and ETCO2 will be recorded as a baseline. Half of the children will be ventilated (with similar values to those of physiologic respiration) and the other half will notThe study is blind, since the anesthesiologist and the dentist would not know if the cuirass of the child is connected to the MRTX or not:

Group 1- 10 children with the cuirass will be connected to the MRTX and artificially ventilated at pressures of (-12/+5) at a rate of 20 per minute, and PO2 and ETCO2 will be recorded every 5 minutes.

Group 2- 10 children with the cuirass will not be connected to the MRTX, but the machine will work at the same condition. Same records of PO2 and ETCO2 will be registered.

DETAILED DESCRIPTION:
The MediventRTX portable lightweight respirator (MRTX) provides noninvasive respiratory support using biphasic extrathoracic ventilation via a cuirass fitted around the patient's chest. The aim of the study is to evaluate the efficacy of the MRTX during dental treatment under deep sedation in comparison with the conventional treatment where children are only under monitor and only intervention is done when required. Twenty healthy children (ASA1) will wear the cuirass. PO2 saturation and ETCO2 will be recorded as a baseline. Half of the children will be ventilated (with similar values to those of physiologic respiration) and the other half will not. The reason of the ventilation is to prevent apnea and high values of PCO2 due to superficial and not efficient breathing. An anesthesiologist is routinely present during treatment under deep sedation. After the child would be deep sedated, he/she will be connected to the cuirass that should be tightly fitted around the patient's chest. The cuirass consists of a clear, flexible plastic enclosure surrounding the chest and abdomen. Its borders are covered by a soft foam rubber, which creates an airtight seal around the patient. By choosing the appropriate cuirass size, the apparatus is capable of ventilating a wide range of different-sized subjects, from infants to the obese adult. The cuirass is connected to a computerized power unit by a wide-bore tube and the respiratory parameters are controlled by a feedback mechanism between the two. The power unit works by creating cyclic pressure changes inside the cuirass. The negative pressure (vacuum) creates chest expansion-inhalation. The positive pressure creates chest compression-exhalation. Thus, both inspiratory and expiratory phases are actively controlled, and the chest is oscillated around a variable negative baseline pressure. The system was found to be effective in a variety of clinical settings, with pressures of -25 to +15 cm H2O, inspiratory/expiratory (I/E) ratios of 1/1 to 1/3, and frequencies of 60 to 150 cpm

The study is blind, since the anesthesiologist and the dentist would not know if the cuirass of the child is connected to the MRTX or not:

Group 1- 10 children with the cuirass will be connected to the MRTX and artificially ventilated at pressures of (-12/+5) at a rate of 20 per minute, and PO2 and ETCO2 will be recorded every 5 minutes.

Group 2- 10 children with the cuirass will not be connected to the MRTX, but the machine will work at the same condition. Same records of PO2 and ETCO2 will be registered.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children (ASA1)
* Need of dental treatment under deep sedation
* Informed consent of parents or guardian

Exclusion Criteria:

* Not healthy children (ASA 2, 3, 4, 5)
* No informed consent

Ages: 12 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2008-07; Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
scores of vital signs with capnograph and pulse oximeter will be recorded at baseline and every five minutes | one session

CONTACTS AND LOCATIONS:
Overall Officials: Diana Ram, DMD, Principal Investigator — Hadassah Medical Organization; David Gozal, MD, Study Chair — Hadassah Medical Organization; Ilan Gur, MD, Study Director — Bikur Holim Hospital
Locations (1):
- Hadassah Medical Organization, Jerusalem, Jerusalem, Israel